CLINICAL TRIAL: NCT03528941
Title: Observational Retrospective Multicenter Study Aimed at Evaluating the Incidence of Hepatitis B Reactivation in Patients Affected by Chronic Lymphocytic Leukemia Treated With Ibrutinib
Brief Title: The Incidence of Hepatitis B Reactivations in Patients Affected by Chronic Lymphocytic Leukemia With Ibrutinib
Acronym: LLC1618
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: LLC1618
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Hepatitis B; Ibrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hepatitis B | interventions — Lamivudine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lamivudine: Patients who received lamivudine
  Interventions: Drug: Lamivudine
- No prophylaxis: Patients who did not receive any prophylaxis
  Interventions: Other: No prophylaxis

INTERVENTIONS:
Drug: Lamivudine — Patients who received lamivudine to prevent hepatitis B
  Groups: Lamivudine
Other: No prophylaxis — Patients who did not receive any prophylaxis to prevent hepatitis B
  Groups: No prophylaxis

SUMMARY:
This observational retrospective study will enroll at least 158 patients affected by Chronic Lymphoid Leukemia (CLL) with previous HBV exposure (HBsAg negative, anti-HBc positive with or without anti-HBs) treated with Ibrutinib single agent according to the IWCLL criteria 2008. Patients will be divided into two cohorts, one encompassing patients who received lamivudine and the second one including patients who received no prophylaxis. Each patient will be observed for one year from the first administration of Ibrutinib.

DETAILED DESCRIPTION:
This observational retrospective study will enroll at least 158 patients affected by CLL with previous HBV exposure (HBsAg negative, anti HBc positive with or without anti-HBs) treated with Ibrutinib single agent according to the IWCLL criteria 2008. Patients will be divided in two cohorts one encompassing patients receiving lamivudine and the second one including patients who will not be given any prophylaxis. Each patient will be observed for one year from the first administration of Ibrutinib.

The aim of the Study is to evaluate the incidence of HBV reactivation cases in patients affected by CLL treated with Ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* CLL/small lymphocytic lymphoma (SLL) patients.
* Patients treated with single-agent Ibrutinib (at least one dose) outside interventional clinical trials before January 31, 2019.
* Serology positive with previous HBV/OBI (HBsAg negatives, anti-HBc positives with or without anti-HBs) infection.
* Signed written informed consent, if applicable, indicating study scope and procedure understanding.

Exclusion Criteria:

* Patients who did not undergo hepatitis B screening before starting the Ibrutinib therapy.
* Patients affected by CLL treated with Ibrutinib vaccinated against hepatitis B or with serology not compatible with a previous infection.
* Patients affected by HCV, HIV or with other causes of liver disease.
* Patients enrolled in clinical trials including Ibrutinib administered in combination with other drugs.
* Patients positive for active hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CLL with previous HBV exposure treated with at least one dose of Ibrutinib.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with hepatitis B reactivation | After 12 months from the first administration of Ibrutinib
  The primary objective of the Study is to evaluate the incidence of HBV reactivation cases in patients affected by CLL treated with Ibrutinib.

SECONDARY OUTCOMES:
Rate of patients managed by prophylaxis | After 12 months from the first administration of Ibrutinib
  number of patients managed by lamivudine prophylaxis
Rate of patients undergoing strict follow-up only | After 12 months from the first administration of Ibrutinib
  number of patients who did not receive any prophylaxis
Rate of HBV reactivation according to patient status and prophylaxis | After 12 months from the first administration of Ibrutinib
  Incidence of HBV reactivation related to patient clinical, biological and therapeutic characteristics, especially in connection with the different incidence of reactivation in patients who received lamivudine prophylaxis versus patients observed with a strict follow-up.
Rate of adverse events during ibrutinib treatment | After 12 months from the first administration of Ibrutinib
  Safety profile in patients who received lamivudine prophylaxis versus patients observed with a strict follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Luca Laurenti, Principal Investigator — Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
Locations (23):
- Italy (23):
  - AOU Arcispedale S.Anna - UOC Ematologia e fisiopatologia della coagulazione, Cona, Ferrara
  - AOU Consorziale Policlinico - UO Ematologia con Trapianto, Bari
  - ASST degli Ospedali Civili di Brescia - UO Ematologia, Brescia
  - AO Brotzu, Presidio Ospedaliero A.Businco - SC Ematologia e CTMO, Cagliari
  - CTC U.O. di Ematologia con Trapianto di midollo osseo - Catania, Catania
  - AO di Catanzaro "Pugliese - Ciaccio", Presidio Ospedaliero "Ciaccio - De Lellis" - Ematologia, Catanzaro
  - Ao Di Cosenza, Presidio Ospedaliero Annunziata - Uoc Ematologia, Cosenza
  - IRCCS AOU San Martino - UO Ematologia e Trapianti, Genova
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Fondazione IRCCS Ca Granda, Ospedale Maggiore Policlinico - Ematologia, Milan
  - IRCCS Ospedale San Raffaele - Unità neoplasie linfocitarie B, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - Fondazione IRCCS Policlinico San Matteo - OU Ematologia, Pavia
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - AOU Pisana - UO Ematologia Universitaria, Pisa
  - AOU Policlinico Tor Vergata - UOC Trapianto cellule staminali, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Area Ematologica, Roma
  - Policlinico Universitario Campus Bio Medico - UOC Ematologia e Trapianto di cellule staminali, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - AOU Città della Salute e della Scienza, Ospedale S.Giovanni Battista Molinette - SC Ematologia, Torino
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it